CLINICAL TRIAL: NCT04466657
Title: A Study to Evaluate Antioxidant Therapy for Moderate to Severe COVID-19 With or Without Comorbidities
Brief Title: Antioxidant Therapy for COVID-19 Study
Acronym: GSHSOD-COVID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Obafemi Awolowo University (Other)
Collaborators: Borno State Ministry of Health (Unknown); Ogun State Ministry of Health (Unknown); Abia State Ministry of Health (Unknown); Sokoto State Ministry of Health (Unknown); Benue State Minsitry of Health (Unknown); University of Calabar Teaching Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GSHSOD-COVID2020
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Covid-19
Keywords: SARS-CoV infection; COVID-19; coronavirus
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Participants in this arm will receive SOC alone, which will be as determined by the clinical team at the treatment centres in line with the current National Interim Guidelines for Clinical Management of COVID-19
  Interventions: Other: Standard of Care
- SOC plus Intervention (Experimental): Participants in this arm will receive SOC plus daily antioxidant supplement composed of two proprietary formulations that include reduced glutathione, N-acetylcysteine, superoxide dismutase, and bovine lactoferrin and immunoglobulins.
  Interventions: Dietary Supplement: Antioxidation Therapy; Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Antioxidation Therapy — Two proprietary formulations composed of reduced glutathione, N-acetylcysteine, superoxide dismutase, and bovine lactoferrin and immunoglobulins.
  Arms: SOC plus Intervention
Other: Standard of Care — SOC will be as determined by the clinical team at the treatment centres in line with the current National Interim Guidelines for Clinical Management of COVID-19

SUMMARY:
Finding effective strategies to treat or prevent the novel coronavirus disease that started in 2019 (COVID-19) is a global public health priority. Potential therapeutics and vaccines are now being investigated in over 1500 clinical trials. Clinical features of the disease include overproduction of reactive oxygen species which induces oxidative stress responses and contribute to acute lung injury. This presents a potential treatment strategy involving antioxidation therapy. In this pilot study, 90 COVID-19 patients aged 18-75 years will be recruited into two groups. The 45 patients in group 1 will receive the standard of care determined by their primary care providers while the 45 patients in group 2 will receive both the standard of care combined with daily antioxidant supplement for 14 days. All patients will be monitored for a total of 28 days with daily monitoring of symptoms and nasopharyngeal swab for SARS-CoV-2 test on days 3, 7, 14 and 28. The study will compare the following between the two groups: (1) the proportion of patients with clinical improvement (defined as live discharge from hospital, decrease of at least 2 points from baseline on a 7-point ordinal scale, or both), and (2) the proportion of patients with negative SARS-CoV-2 test by PCR on days 3, 7, and 14.

DETAILED DESCRIPTION:
Background: COVID-19 caused by SARS-CoV-2 is an unprecedented global public health challenge which as at 06 May 2020 has spread to over 210 with over 3.6 million cases including 250,000 deaths. More than 1500 clinical trials are currently ongoing in an unprecedented global search for potential therapeutics and vaccines. Certain clinical features of SARS-CoV-2 infection provide potential treatment strategies involving antioxidation therapy, including overproduction of reactive oxygen species which induces oxidative stress responses and contribute to acute lung injury.

Primary Outcome Measure: (1) the proportion of patients with clinical improvement (defined as live discharge from hospital, decrease of at least 2 points from baseline on a 7-point ordinal scale, or both), and (2) the proportion of patients with negative SARS-CoV-2 test by PCR on days 3, 7, and 14.

Study Design: Individuals within 18-75 years of age who receive a PCR positive test for COVID-19 and admitted at participating COVID-19 isolation and treatment centres will be invited to participate. Consenting individuals will be randomised 1:1 to receive either standard of care alone (control group) or standard of care plus daily antioxidant supplementation (intervention group). A total of 90 participants will be recruited in the Pilot Stage (n = 45 per arm). The Pivotal Stage will include 300 participants. Antioxidant therapy will be a formulation composed of reduced GSH, N-acetylcysteine, superoxide dismutase and bovine lactoferrin and immunoglobulin as in whey protein isolate. Clinical improvement will be evaluated daily using a 7-category ordinal scale. SARS-CoV-2 PCR test will be repeated on days 3, 7, 14 and 28.

Analysis: An interim analysis of data from the Pilot Stage will be conducted after the first 45 participants have completed days 1-14 of the study period. These data will provide valuable insights regarding possible revision of the design, conduct and analysis of the Pivotal Stage. Analysis of clinical improvement based on the 7-category ordinal scale will be performed using time-to-event data (patients will censored at 28-days of follow-up). Categorical variables will be analysed using the log-rank test and continuous variables will be assessed using a univariable Cox proportional hazard regression analysis. Proportion of participants with SARS-CoV-2 polymerase chain reaction (PCR) negative result at days 3, 7, 14 and 28 will be compared between the intervention and control groups.

Ethics: This trial will be conducted in compliance with the protocol, the principles of ICH Guideline E6 for Good Clinical Practice, the Declaration of Helsinki, and all applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent prior to any study procedures
* Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test ≤ 2 days before randomization
* Currently hospitalized and requiring medical care for COVID-19
* Peripheral capillary oxygen saturation (SpO2) < 94% on room air at screening

Exclusion Criteria

* Participation in any other clinical trial of an experimental treatment for COVID-19
* Concurrent treatment with other agents outside the standard of care than 24 hours prior to study intervention dosing
* Requiring mechanical ventilation at screening
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) above 5 times upper limit of normal (ULN)
* Creatinine clearance < 50 mL/min using the Cockcroft-Gault formula

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | 28 days
  Time to clinical improvement (defined as time from randomization to either an improvement of two points on a 7-category ordinal scale or discharge from the hospital, whichever came first, or both)
Time to SARS-CoV-2 negativity | 14 days
  Proportion of participants with SARS-CoV-2 polymerase chain reaction (PCR) negative result at Day 14

SECONDARY OUTCOMES:
Clinical status on day 14 | 14 days
  Clinical status as assessed with the seven-category ordinal scale on day 14
Proportion of participants with SARS-CoV-2 PCR negative result at Day 7 | 7 days
Proportion of participants with SARS-CoV-2 PCR negative result at Day 28 | 28 days
28 Day mortality | 28 days
Duration of hospitalization in survivors | 28 days
Time from treatment initiation to death | 28 days

OTHER OUTCOMES:
Adverse events during treatment | 28 days
Serious adverse events | 28 days
  Respiratory failure or Acute Respiratory Distress Syndrome, Acute Kidney Injury, secondary infection, shock, severe anemia, acute gastritis, unconsciousness, acute heart failure
Gastrointesntinal adverse events | 28 days
  Nausea, vomiting, and diarrhea
Discontinuation of trial intervention before the end of protocol specified 14 days | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Adeniyi Olagunju, BPharm, MRes, PhD, Study Chair — Obafemi Awolowo University
Locations (11):
- Nigeria (11):
  - Abia State Isolation Centre, Amachara, Umuahia, Abia State
  - Benue State University Teaching Hospital, Makurdi, Benue State
  - Brigadier Abba Kyari Memorial Hospital, Borno, Borno State
  - University of Maiduguri Teaching Hospital, Maiduguri, Borno State
  - University of Calabar Teaching Hospital, Calabar, Cross River State
  - Federal Medical Centre Idi-Aba, Abeokuta, Ogun State
  - Olabisi Onabanjo University Teaching Hospital, Sagamu, Ogun State
  - Infectious Disease Hospital, Ammanawa, Sokoto State
  - Murtala Muhammad Speciaist Hospital, Sokoto, Sokoto State
  - Occupational Therapy Center, Sokoto, Sokoto State
  - Usmanu Danfodiyo University Teaching Hospital, Sokoto, Sokoto State

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuki K, Fujiogi M, Koutsogiannaki S. COVID-19 pathophysiology: A review. Clin Immunol. 2020 Jun;215:108427. doi: 10.1016/j.clim.2020.108427. Epub 2020 Apr 20. PMID 32325252
- [Background] Imai Y, Kuba K, Neely GG, Yaghubian-Malhami R, Perkmann T, van Loo G, Ermolaeva M, Veldhuizen R, Leung YH, Wang H, Liu H, Sun Y, Pasparakis M, Kopf M, Mech C, Bavari S, Peiris JS, Slutsky AS, Akira S, Hultqvist M, Holmdahl R, Nicholls J, Jiang C, Binder CJ, Penninger JM. Identification of oxidative stress and Toll-like receptor 4 signaling as a key pathway of acute lung injury. Cell. 2008 Apr 18;133(2):235-49. doi: 10.1016/j.cell.2008.02.043. PMID 18423196
- [Background] Hosakote YM, Jantzi PD, Esham DL, Spratt H, Kurosky A, Casola A, Garofalo RP. Viral-mediated inhibition of antioxidant enzymes contributes to the pathogenesis of severe respiratory syncytial virus bronchiolitis. Am J Respir Crit Care Med. 2011 Jun 1;183(11):1550-60. doi: 10.1164/rccm.201010-1755OC. Epub 2011 Mar 4. PMID 21471094
- [Background] Lin X, Wang R, Zou W, Sun X, Liu X, Zhao L, Wang S, Jin M. The Influenza Virus H5N1 Infection Can Induce ROS Production for Viral Replication and Host Cell Death in A549 Cells Modulated by Human Cu/Zn Superoxide Dismutase (SOD1) Overexpression. Viruses. 2016 Jan 8;8(1):13. doi: 10.3390/v8010013. PMID 26761025
- [Background] Cao W, Liu X, Bai T, Fan H, Hong K, Song H, Han Y, Lin L, Ruan L, Li T. High-Dose Intravenous Immunoglobulin as a Therapeutic Option for Deteriorating Patients With Coronavirus Disease 2019. Open Forum Infect Dis. 2020 Mar 21;7(3):ofaa102. doi: 10.1093/ofid/ofaa102. eCollection 2020 Mar. PMID 32258207
- [Background] Sinha R, Sinha I, Calcagnotto A, Trushin N, Haley JS, Schell TD, Richie JP Jr. Oral supplementation with liposomal glutathione elevates body stores of glutathione and markers of immune function. Eur J Clin Nutr. 2018 Jan;72(1):105-111. doi: 10.1038/ejcn.2017.132. Epub 2017 Aug 30. PMID 28853742